CLINICAL TRIAL: NCT00234754
Title: Surgical Management of Stress Urinary Incontinence in Women: A Randomized Clinical Trial (RCT) of TOT vs TVT
Brief Title: Trans-Obturator Tape Versus Trans-Vaginal Tape for Stress Urinary Incontinence in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Health services (Other); Boston Scientific Corporation (Industry); Alberta Heritage Foundation for Medical Research (Other)
Responsible Party: Principal Investigator, Dr. Sue Ross, Adjunct Professor, Obstetrics and Gynecology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18421; 200400964
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Stress Urinary Incontinence
Keywords: Incontinence; Surgery; Trans-vaginal tape; Trans-obturator tape
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Trans-vaginal tape Surgery
  Interventions: Procedure: TVT Surgery TOT Surgery
- 2 (Experimental): Trans-obturator tape surgery
  Interventions: Procedure: TVT Surgery TOT Surgery

INTERVENTIONS:
Procedure: TVT Surgery TOT Surgery — TVT surgery and TOT surgery

SUMMARY:
Stress urinary incontinence (SUI) is a health concern for many women. The transvaginal tape (TVT) surgery has become a common procedure to address the problem. Another surgery is now available, trans-obturator tape (TOT). The investigators will compare these 2 approaches to dealing with SUI and follow the women for 1 year. Women will also be followed at 5 years after surgery.

DETAILED DESCRIPTION:
This study is a randomized trial in which women with stress incontinence will be allocated to receive either TOT or TVT procedures. Women who elect surgical management of their type II stress incontinence are eligible to participate in the trial. Baseline data, including a patient questionnaire, will be collected. Hospital outcomes, including length of stay and surgical complications will be documented from hospital charts. All women attend a 6-week follow-up visit as standard of care: a structured data collection form will be used by surgeons to collect information and another patient questionnaire will be administered. At 12 months postoperatively women will attend the clinic for objective measurement of incontinence, a full exam and to complete a questionnaire. The main outcome is effectiveness of the procedure determined using a 1-hour pad test. Secondary research questions include:

How effective is TOT compared to TVT in terms of:

Subjective cure at 12 months postoperatively? Incontinence-specific quality of life at 6 weeks and 12 months postoperatively? Satisfaction with surgery at 12 months postoperatively? Return to usual activities and usual sex life after surgery? The prevalence of voiding dysfunction at 12 months postoperatively? Surgical complications, both short term and long term? Utility and cost? (an economic evaluation) The study will be carried out according to the ICH Good Clinical Practice Guidelines.

At 5 years postoperatively women will attend the clinic for a further follow-up. The primary research question of the 5-year follow-up is:

Safety - What is the incidence of vaginal erosion or other serious adverse outcomes of surgery among women who had a surgical procedure for stress urinary incontinence utilizing a TOT device, versus a TVT device, over the 5 years following surgery?

Secondary questions are as follows:

Effectiveness - What are the objective and subjective outcomes of TOT compared with TVT at 5 years following surgery for SUI? Health economics - What are the disease-specific rates of health service utilization related to repeat surgical intervention, as well as surgery and other treatment related to adverse events for women who had a TOT procedure, versus those who had a TVT procedure, over the 5 years after surgery? Using economic modelling and cost utility analysis, is TOT cost-effective compared with TVT over the 5 years after surgery?

Other question:

Do women with tape found to be palpable in the vagina at 12 months postoperatively, go on to develop vaginal erosion by 5 years following surgery?

ELIGIBILITY:
Inclusion Criteria:

* Women with type II stress incontinence, defined as leaking with increased abdominal pressure
* Are eligible for both types of surgery

Exclusion Criteria:

* Have vaginal prolapse requiring surgical repair
* Have had previous incontinence surgery
* Have overactive bladder or incontinence is caused only by bladder overflow
* Intend to have further children
* Have Alzheimer's or Parkinson's disease, progressive neurological disease such as multiple sclerosis, or are immunocompromised
* Are unable to understand English
* Will be unavailable for follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2005-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
How effective is TOT compared to TVT in terms of objective cure at 12 months postoperatively? | 1 year
  Objective evidence of SUI will be obtained using a standardised pad test undertaken at 12 months following surgery. The pad test will be carried out using a modification of the International Continence Society (ICS) recommendations. Women will be considered 'cured' if the pad weight gain is less than 1g over the test period. This is the definition of cure used by Ward and will allow comparison with that trial.
Vaginal erosion or other serious adverse outcomes of surgery over 5 years postoperatively | 5 years

SECONDARY OUTCOMES:
How effective is TOT compared to TVT in terms of subjective cure 12 months postoperatively? | 1 year
Incontinence-specific quality of life at 6 weeks and 12 months postoperatively? | 1 year
Satisfaction with surgery at 12 months postoperatively? | 1 year
Return to usual activities and usual sex life after surgery? | 6 weeks and 1 year
The prevalence of voiding dysfunction at 12 months postoperatively? | 1 year
Surgical complications, both short term and long term? | 6 weeks and 1 year
Utility and cost? (an economic evaluation) | 1 year
Subjective effectiveness at 5 years postoperatively | 5 years
Incontinence-specific quality of life at 5 years postoperatively | 5 years
  Urogenital Distress Inventory (UDI-6), Incontinence Impact Questionnaire (IIQ-7, Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12)
Health care utilization over 5 years postoperatively | 5 year
Cost effectiveness over 5 years postoperatively | 5 year
Objective effectiveness at 5 years postoperatively | 5 years
  Pad test leakage of <1g over period of test

CONTACTS AND LOCATIONS:
Overall Officials: Sue Ross, PhD, Principal Investigator — University of Calgary; Magali Robert, MD, Principal Investigator — Univerty of Calgary, Calgary Health Region
Locations (1):
- Calgary Health Region, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Decision to share will depend on review of IPD protocol

REFERENCES:
- [Background] Ross S, Robert M, Lier D, Eliasziw M, Jacobs P. Surgical management of stress urinary incontinence in women: safety, effectiveness and cost-utility of trans-obturator tape (TOT) versus tension-free vaginal tape (TVT) five years after a randomized surgical trial. BMC Womens Health. 2011 Jul 22;11:34. doi: 10.1186/1472-6874-11-34. PMID 21781314
- [Result] Ross S, Robert M, Swaby C, Dederer L, Lier D, Tang S, Brasher P, Birch C, Cenaiko D, Mainprize T, Murphy M, Carlson K, Baverstock R, Jacobs P, Williamson T. Transobturator tape compared with tension-free vaginal tape for stress incontinence: a randomized controlled trial. Obstet Gynecol. 2009 Dec;114(6):1287-1294. doi: 10.1097/AOG.0b013e3181c2a151. PMID 19935032
- [Result] Lier D, Ross S, Tang S, Robert M, Jacobs P; Calgary Women's Pelvic Health Research Group. Trans-obturator tape compared with tension-free vaginal tape in the surgical treatment of stress urinary incontinence: a cost utility analysis. BJOG. 2011 Apr;118(5):550-6. doi: 10.1111/j.1471-0528.2010.02845.x. Epub 2011 Feb 4. PMID 21291510
- [Result] Ross S, Tang S, Eliasziw M, Lier D, Girard I, Brennand E, Dederer L, Jacobs P, Robert M. Transobturator tape versus retropubic tension-free vaginal tape for stress urinary incontinence: 5-year safety and effectiveness outcomes following a randomised trial. Int Urogynecol J. 2016 Jun;27(6):879-86. doi: 10.1007/s00192-015-2902-7. Epub 2015 Dec 15. PMID 26670575
- [Result] Lier D, Robert M, Tang S, Ross S. Surgical treatment of stress urinary incontinence-trans-obturator tape compared with tension-free vaginal tape-5-year follow up: an economic evaluation. BJOG. 2017 Aug;124(9):1431-1439. doi: 10.1111/1471-0528.14227. Epub 2016 Aug 10. PMID 27506185